CLINICAL TRIAL: NCT04268563
Title: Comparing the Therapeutic Effect of Sitagliptin/Metformin and Metformin on Biochemical Factors and Expression of GDF-9 and BMP-15 Genes in Patients With Classic PCOS Undergoing Intra-cytoplasmic Sperm Injection (ICSI)
Brief Title: Comparing the Effect of Sitagliptin/Metformin and Metformin in PCOS Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Delbar Daneshjou, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11367
Record Dates: First submitted 2020-01-28; First posted 2020-02-13 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Polycystic Ovary Syndrome; Infertility; ART
Keywords: metformin; sitagliptin; Polycystic Ovary Syndrome; Intracytoplastic sperm injection
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Rehydration Solutions; Metformin; Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Control group: oral rehydration salts (ORS, Poursina, Tehran, Iran), two times daily
  Interventions: Drug: placebo
- Metformin (Experimental): Intervention group 1: received Metformin (Glucophage, Merck, West Drayton, UK; 500 mg ,two times daily
  Interventions: Drug: metformin
- Sitagliptin (Experimental): Intervention group2: received Sitagliptin (Januvia, Merck,West Drayton, UK. 50 mg, two times daily
  Interventions: Drug: Sitagliptin
- sitagliptin/metformin (Experimental): Intervention group3: received Sitagliptin/metformin (Janumet, Merck,West Drayton, UK. 50/500 mg), two times daily
  Interventions: Drug: Sitagliptin/metformin

INTERVENTIONS:
Drug: placebo — Oral rehydration solution
  Other Names: rehydration solution
  Arms: Placebo
Drug: metformin — metformin tablet
  Other Names: Glucophage
  Arms: Metformin
Drug: Sitagliptin — Sitagliptin tablet
  Other Names: JANUVIA
  Arms: Sitagliptin
Drug: Sitagliptin/metformin — Sitagliptin/metformin tablet
  Other Names: JANUMET
  Arms: sitagliptin/metformin

SUMMARY:
Investigators will evaluate and compare the efficacy of Sitagliptin/Metformin to metformin and sitagliptin on gdf9 and bmp15 gene expression on PCOS patients undergoing intracytoplasmic sperm injection(ICSI).

DETAILED DESCRIPTION:
This study was conducted in Infertility clinic of Mahdiyeh Educational Hospital, Tehran. Patients in the four groups receive the drug 2 months before the start of the ovulation cycle, and treatment will continue until the day of the oocyte aspiration. The drug provide by midwife to patients and both patient and physician blind to the treatment regimen. The participants randomly divide into four groups.The ovulation induction stimulate with GnRh antagonist.

ELIGIBILITY:
Inclusion Criteria:

* subject has clinical or biochemical hyperandrogenic symptoms
* subject has oligo/amenorrhea cycles

Exclusion Criteria:

* Hypersensitivity to metformin
* Hypersensitivity to sitagliptin presence of infertility factors other than anovulation,
* male infertility
* pelvic organic pathologies
* congenital adrenal hyperplasia
* thyroid dysfunction
* Cushing's syndrome
* hyper prolactinemia
* androgen secreting neoplasia
* diabetes mellitus
* consumption of medications affecting carbohydrate metabolism
* consumption hormonal analogues other than progesterone 2 months prior to enrolment in the study
* severe hepatic
* pancreatitis
* kidney diseases
* gallbladder diseases

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study is based women with polycystic ovary syndrome.
Enrollment: 80 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-07-19 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Fasting insulin | 24 hours after last dose
  ELIZA hormone assay
Growth differentiation factor-9(GDF-9) expression | 24 hours after last dose
  Realtime PCR
Bone morphogenetic protein-15(BMP-15) expression | 24 hours after last dose
  Realtime PCR
Total Testosterone | 24 hours after last dose
  ELIZA hormone assay
Follicle-stimulating hormone(FSH) | 24 hours after last dose
  ELIZA hormone assay

CONTACTS AND LOCATIONS:
Overall Officials: Shahrzad Shahrzad Zadehmodarres, Professor, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Mahdiyeh educational hospital, Tehran, Iran

REFERENCES:
- [Derived] Daneshjou D, Zadeh Modarres S, Soleimani Mehranjani M, Shariat Zadeh SMA. Comparing the effect of sitagliptin and metformin on the oocyte and embryo quality in classic PCOS patients undergoing ICSI. Ir J Med Sci. 2021 May;190(2):685-692. doi: 10.1007/s11845-020-02320-5. Epub 2020 Jul 28. PMID 32720198